CLINICAL TRIAL: NCT02522624
Title: Supporting Decisions About Health Insurance to Improve Care for the Uninsured
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201407058; 5R01MD008808-02 (NIH)
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Health Literacy; Health Insurance; Health Services Accessibility; Informed Decision Making
Keywords: Health insurance; Health services accessibility; Decision making; Health literacy
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decision Aid (DA) (Experimental): The decision aid (DA) will be provided to participants randomized to the experimental/intervention group.
  Interventions: Behavioral: Decision Aid (DA)
- Control (No Intervention): Participants randomized to the control group will receive usual care. They will be directed to the healthcare.gov website and asked to follow the prompts to view and select (if applicable) a health insurance plan.

INTERVENTIONS:
Behavioral: Decision Aid (DA) — Participants will be shown (on a computer) a targeted, web-based decision aid focused on the topic of health insurance plans in addition to usual care.
  Arms: Decision Aid (DA)

SUMMARY:
The overall purpose of the study is to better understand how the investigators previously developed decision support (DS) tool can help people make decisions about health insurance plans available through the federal exchanges created by the Affordable Care Act (ACA). The investigators will evaluate the DS tool compared to the federal government website. The investigators will also evaluate the feasibility of disseminating this tool. There are two primary aims to be completed in this project: (1) examine the reach and effectiveness of the health insurance DS tool; and (2) collect stakeholders' feedback to improve the likelihood of implementation of the DS tool.

DETAILED DESCRIPTION:
First, for Aim 1 part 1, the investigators will recruit 40 key stakeholders (uninsured participants, health providers, community advisors, and health policy experts) to refine the DS tool through a series of individual semi-structured interviews. Next, the investigators will use their feedback to program the DS strategies into an online DS tool. After its initial production, the tool will be pilot tested with 30 individuals to assess readability, message clarity, format, and function of the tool as well as to test the randomized trial study procedures. Then, for Aim 1 part 2, the investigators will test the DS tool in a randomized trial with 362 participants eligible for the Affordable Care Act (ACA) exchanges. Half will use the DS tool and the other half will use the federal government site to learn about the exchanges. The investigators will use computerized random assignment to assign participants to study condition, after which they will all complete the same short survey. For Aim 2, the investigators will collect 40 stakeholders' feedback on likelihood of adoption and implementation of the DS tool to plan for dissemination and implementation. Stakeholders will be asked both open-ended and closed-ended questions in order to gather feedback about delivering the DS tool. These stakeholders will be different from those who were interviewed in Aim 1 as to ensure broader applicability of the DS tool.

ELIGIBILITY:
Inclusion Criteria:

* Must be without health insurance currently; or
* Must be enrolled in one of the ACA exchange plans in the past 1 year; and
* Must speak English

Exclusion Criteria:

* Currently has health insurance that was not provided by being enrolled in one of the ACA exchange plans in the past year
* Currently has health insurance that is provided through public insurance or private employer-based insurance
* Does not speak English

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 328 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Politi, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- The Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Politi MC, Barker AR, Kaphingst KA, McBride T, Shacham E, Kebodeaux CS. Show Me My Health Plans: a study protocol of a randomized trial testing a decision support tool for the federal health insurance marketplace in Missouri. BMC Health Serv Res. 2016 Feb 16;16:55. doi: 10.1186/s12913-016-1314-9. PMID 26880251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 10/2015 - 1/2016 via community events, online advertisements, social service organizations, and the recruitment/retention arm of our Center for Community-Engaged Research.
Pre-assignment Details: 482 participants were assessed for eligibility. Participants were excluded (n=154) if they did not meet the inclusion criteria (n=82) or could not be reached (n=65).
Period: Overall Study
Arm/Group | Decision Aid (DA) | Control
Started | 165 | 163
Completed | 164 (Discontinued intervention due to technical failure (n=1)) | 163
Not Completed | 1 | 0
Not completed — Technical failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid (DA) | Control | Total
Number analyzed (Participants) | 164 | 163 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (13.2) | 41.4 (12.5) | 42.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 94 | 191
  Male | 67 | 69 | 136
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic | 156 | 159 | 315
  Hispanic | 8 | 4 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  African American only | 96 | 107 | 203
  Caucasian only | 46 | 41 | 87
  Other (Including Mixed) | 22 | 15 | 37
Education [Number; unit: participants]
  Less than HS | 12 | 15 | 27
  HS or GED | 111 | 99 | 210
  College + | 41 | 49 | 90
% Federal Poverty Line [Number; unit: participants] — Four participants in the healthcare.gov condition did not report FPL (n=159)
  participants
    < 100 | 72 | 94 | 166
    100-249 | 64 | 47 | 111
    250-399 | 15 | 10 | 25
    400+ | 13 | 8 | 21
Urbanicity [Number; unit: participants]
  Rural | 9 | 11 | 20
  Suburban | 97 | 99 | 196
  Urban | 58 | 53 | 111
Total number covering [Number; unit: participants]
  1 | 97 | 106 | 203
  2 | 32 | 21 | 53
  3+ | 35 | 36 | 71
Smoking status - Participant [Number; unit: participants]
  Yes | 55 | 47 | 102
  No | 109 | 116 | 225
Smoking status - Dependent (n=124) [Number; unit: participants] — n=124
  participants
    Yes | 10 | 9 | 19
    No | 57 | 48 | 105
Chronic Conditions - Participant (n=207) [Mean (Standard Deviation); unit: Number chronic conditions] — Population: Only participants specifying they have a chronic condition were asked to provide the number of chronic conditions.
  Number chronic conditions
    number analyzed (Participants) | 96 | 111 | 207
    (all) | 2.27 (1.53) | 2.17 (1.35) | 2.22 (1.43)
Chronic Conditions - Participant + Dependents (n=107) [Mean (Standard Deviation); unit: Number chronic conditions] — Population: Only participants with dependents were asked to provide the number of chronic conditions anyone in their household had (if any).
  Number chronic conditions
    number analyzed (Participants) | 107 | 163 | 270
    (all) | 2.69 (2.35) | NA (NA) — Participants in Control condition were not asked about their dependents' chronic conditions. | NA (NA) — Only participants in the DA group were asked about their dependents' chronic conditions to allow the DA tool to personalize good fit plans.
Insurance Status (Uninsured) [Number; unit: participants]
  Uninsured | 85 | 93 | 178
  Insured | 79 | 70 | 149
Health Literacy (SILS) [Number; unit: participants] — The Single Item Literacy Screener (SILS) assessed broader health literacy. The SILS is a single item question intended to identify adults in need of help with printed health material scored on a scale from 1-5 (1 indicating never needing help with printed health material; 5 indicating always needing help with printed health material). Participants with scores greater than 2 were categorized into the "limited" health literacy category; remaining participants were categorized into "adequate" category.
  One participant in the healthcare.gov condition did not complete the SNS or SILS (n=162)
  participants
    Adequate | 139 | 128 | 267
    Limited | 25 | 34 | 59
Subjective Numeracy (SNS) [Mean (Full Range); unit: units on a scale] — Three items from the Subjective Numeracy Scale (SNS) assessed numeracy skills. The SNS is a self-report measure scored from 1-6, with larger values indicating greater perceived ability with mathematical tasks. Scores from each of the three items were summed and averaged to obtain a composite score. Values for Range are the actual score range obtained from the study's participants.
  One participant in the healthcare.gov condition did not complete the SNS or SILS (n=162)
  units on a scale | 3.9 [1 to 6] | 3.6 [1 to 6] | 3.8 [1 to 6]
Objective Numeracy (Lipkus) [Mean (Full Range); unit: units on a scale] — Four items from a validated objective numeracy scale assessed numeracy skills. Each of the open-ended responses to the four items were scored correct or incorrect. The number of correct items were summed to obtain a summary score. Values for Range are the actual score range obtained from the study's participants.The mean of the summary score was obtained to provide average scores for the DA and Control groups.
  units on a scale | 2.6 [0 to 4] | 2.3 [0 to 4] | 2.4 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Score (% Correct)
Description: 8 questions developed in researchers' past work. Assessed health insurance knowledge.
Time Frame: Completed immediately after reviewing Decision Aid tool, taking about 5 minutes to complete.
Measure: Mean (Standard Deviation); unit: percentage of 8 items correctly answered
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 164 | 163
percentage of 8 items correctly answered | 77.6 (18.2) | 58.8 (21.0)
Statistical Analysis 1: Comparison: Decision Aid (DA) vs Control; Test type: Superiority or Other; p < .001, Regression, Linear — A priori sample size estimates yielded an estimate of 183 per group needed to detect an effect size of 0.34 with 90% power at a 0.05 level of significance and 137 per group with 80% power
Statistical Analysis 2: Comparison: Decision Aid (DA) vs Control; Examined the relation between group and categorical outcomes, controlling for % Federal Poverty Level (400 or greater, 250-399, 100-249, less than 100); Test type: Superiority or Other; p = 0.16, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Aid (DA) vs Control; Controlling for Numeracy; Test type: Superiority or Other; p < .001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Decision Self-efficacy
Description: The decision self-efficacy (DSE) scale measured participants' perceived ability to understand insurance info and resist unwanted decision pressure. The 6 items on the DSE scale were each rated on a 3-point scale (0=Not confident; 2=A little confident; 4=Very confident). The sum of the DSE items was divided by 6 and multiplied by 25 to obtain a score on a 0-100 scale. Higher values indicate more confidence in one's decision-making ability.
Time Frame: Completed immediately after reviewing Decision Aid tool, taking about 5 minutes to complete.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 164 | 163
units on a scale | 81.5 (22.5) | 73.0 (20.4)
Statistical Analysis 1: Comparison: Decision Aid (DA) vs Control; Test type: Superiority or Other; p = 0.002, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Aid (DA) vs Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.30, Regression, Linear
Statistical Analysis 3: Comparison: Decision Aid (DA) vs Control; Controlling for Numeracy; Test type: Superiority or Other; p = 0.82, Regression, Linear

3. Primary Outcome: Confidence in Choice
Description: The 4-item SURE (Sure of myself; Understand information; Risk-benefit ratio; Encouragement) decisional conflict scale assessed confidence in plan choice. Each item could be answered dichotomously (1=yes; 0=no). Responses were summed and a group average was obtained. Higher SURE values indicate more confidence in choice. The scale ranged from 0-4.
Time Frame: Completed immediately after reviewing Decision Aid tool, taking about 5 minutes to complete.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 164 | 163
units on a scale | 3.5 (0.9) | 2.9 (1.3)
Statistical Analysis 1: Comparison: Decision Aid (DA) vs Control; Test type: Superiority or Other; p < .001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Aid (DA) vs Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.82, Regression, Linear
Statistical Analysis 3: Comparison: Decision Aid (DA) vs Control; Controlling for Numeracy; Test type: Superiority or Other; p = 0.15, Regression, Linear

4. Secondary Outcome: Improvements in HILM 1 (Health Insurance Literacy Measure)
Description: Assessed confidence estimating costs of care.Improvement in HILM was defined as moving from "not confident" pre-intervention to "a little confident" or "very confident" post-intervention, or from "a little confident" pre-intervention to "very confident" post-intervention.
Time Frame: Pre-intervention and post-intervention
Population: One participant in healthcare.gov (Control) condition did not finish HILM (n=162)
Measure: Number; unit: participants
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 164 | 162
participants
  Yes | 66 | 49
  No | 98 | 113
Statistical Analysis 1: Comparison: Decision Aid (DA) vs Control; Test type: Superiority or Other; p = 0.10, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.92 to 2.36]
Statistical Analysis 2: Comparison: Decision Aid (DA) vs Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.26, Regression, Logistic
Statistical Analysis 3: Comparison: Decision Aid (DA) vs Control; Controlling for Numeracy; Test type: Superiority or Other; p = 0.58, Regression, Linear

5. Secondary Outcome: Improvements in HILM 2 (Health Insurance Literacy Measure)
Description: Assessed confidence understanding terms.Improvement in HILM was defined as moving from "not confident" pre-intervention to "a little confident" or "very confident" post-intervention, or from "a little confident" pre-intervention to "very confident" post-intervention.
Time Frame: Pre-intervention and post-intervention
Population: One participant in healthcare.gov (Control) condition did not finish HILM (n=162)
Measure: Number; unit: participants
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 164 | 162
participants
  Yes | 88 | 51
  No | 76 | 111
Statistical Analysis 1: Comparison: Decision Aid (DA) vs Control; Test type: Superiority or Other; p < .001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.52, 95% CI 2-sided [1.58 to 4.01]
Statistical Analysis 2: Comparison: Decision Aid (DA) vs Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.39, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Aid (DA) vs Control; Controlling for Numeracy; Test type: Superiority or Other; p = 0.57, Regression, Linear

6. Secondary Outcome: Intended Choice Metal Level
Description: Participants indicated the plan they would choose that day. We categorized plans by governmental classifications of metal level (catastrophic, bronze, silver, gold).
Time Frame: Completed immediately after reviewing Decision Aid tool, taking about 5 minutes to complete.
Population: Intended plan choice metal level data were not available for 2 participants in SMHP (Show Me My Health Plans decision aid) condition (n=162) and for 11 participants in healthcare.gov (Control) condition (n=152)
Measure: Number; unit: participants
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 162 | 152
participants
  Catastrophic | 0 | 5
  Bronze | 41 | 108
  Silver | 121 | 30
  Gold | 0 | 9
  Platinum | 0 | 0
Statistical Analysis 1: Comparison: Decision Aid (DA) vs Control; Test type: Superiority or Other; p < .001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 10.32, 95% CI 2-sided [5.94 to 17.95]
Statistical Analysis 2: Comparison: Decision Aid (DA) vs Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Aid (DA) vs Control; Controlling for numeracy; Test type: Superiority or Other; p = 0.46, Regression, Linear

ADVERSE EVENTS:
Arm/Group | Decision Aid (DA) | Control
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/163
Other Adverse Events (participants affected / at risk) | 0/165 | 0/163

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No